CLINICAL TRIAL: NCT00141687
Title: Early External Cephalic Version 2 Trial
Brief Title: Early External Cephalic Version (ECV) 2 Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of British Columbia (Other)
Responsible Party: Principal Investigator, Eileen Hutton, Professor, Department of Obstetrics & Gynecology, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C04-0348; ISRCTN56498577
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Breech Presentation
Keywords: External cephalic version; Cesarean section; pregnancy; labour; Breech pregnancy
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early External Cephalic Version Group (Experimental): Early external cephalic version (ECV) procedure performed between 34 weeks and 0/7 days and 35 weeks and 6/7 days of gestation
  Interventions: Procedure: Early ECV between 34 0/7 and 35 6/7 weeks
- Delayed External Cephalic Version Group (Active Comparator): Delayed external cephalic version (ECV) procedure performed at or after 37 weeks and 0/7 days of gestation
  Interventions: Procedure: Delayed ECV at or after 37 0/7 weeks

INTERVENTIONS:
Procedure: Early ECV between 34 0/7 and 35 6/7 weeks — Early external cephalic version between 34 0/7 and 35 6/7 weeks of gestation
  Other Names: Early External Cephalic Version (ECV)
  Arms: Early External Cephalic Version Group
Procedure: Delayed ECV at or after 37 0/7 weeks — Delayed external cephalic version at or after 37 0/7 weeks of gestation
  Other Names: Delayed External Cephalic Version (ECV)
  Arms: Delayed External Cephalic Version Group

SUMMARY:
For women with a fetus in breech presentation, does early ECV (at 34 0/7 up to 35 weeks and 6/7 days) versus delayed ECV (not before 37 weeks and 0/7 days) increase or decrease the likelihood of cesarean section (CS)?

DETAILED DESCRIPTION:
Primary Outcomes: Rate of Caesarean section

Secondary Outcomes: Rate of preterm birth

Other Outcomes: admission to neonatal intensive care unit ≥ 24 hours, perinatal or neonatal mortality or serious neonatal morbidity, serious fetal complications, maternal death or serious maternal morbidity, non-cephalic presentation at birth, women's views, and health care costs.

The Data Coordination for this study is being carried out at the Maternal, Infant Reproductive Health Research Unit at Sunnybrook and Women's College Health Sciences Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Women with any breech presentation
2. A live singleton fetus
3. Gestational age of 33 weeks 0 days to 35 weeks 6 days

Exclusion Criteria:

1. Contraindications to ECV (e.g. fetal heart rate abnormalities, abruptio placenta, major life-threatening fetal anomalies, uterine anomalies, hyper-extended fetal head, rupture of membranes, severe oligohydramnios, severe polyhydramnios)
2. Contraindications to early ECV (e.g. increased risk of preterm labour [such as past history of preterm labour in this or previous pregnancies], increased risk of abruptio placenta [such as maternal hypertension])
3. Contraindications to labour or vaginal delivery (e.g. placenta previa, previous classical CS)
4. Women planning delivery by CS if the fetus turns to cephalic
5. Women planning a vaginal delivery if the fetus remains breech
6. Women at increased risk of unstable lie (eg. grand multiparity)
7. Previous participation in EECV2 Trial

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1543 (Actual)
Dates: Start 2004-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Rate of cesarean section | Information not available

SECONDARY OUTCOMES:
Rate of pre-term births. Other outcomes: admission to neonatal intensive care unit ≥ 24 hours, perinatal or neonatal mortality or serious neonatal morbidity, or others. | Information not available

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Eileen Hutton, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- See also: Main results: Hutton EK et al. The Early External Cephalic Version (ECV) 2 Trial: an international multicentre randomised controlled trial of timing of ECV for breech pregnancies. BJOG. 2011 Apr;118(5):564-77. — http://www.ncbi.nlm.nih.gov/pubmed/21291506
- See also: Reitsma A et al. Accounting for center in the Early External Cephalic Version trials: an empirical comparison of statistical methods to adjust for center in a multicenter trial with binary outcomes. Trials. 2014 Sep 26;15:377. — http://www.ncbi.nlm.nih.gov/pubmed/25257928
- See also: Murray-Davis B. et al. Women's experiences of participating in the early external cephalic version 2 trial. Birth. 2012 Mar;39(1):30-8 — http://www.ncbi.nlm.nih.gov/pubmed/22369603
- See also: Cost analysis: Ahmed RJ, Gafni A, Hutton EK. The Cost Implications in Ontario, Alberta, and British Columbia of Early Versus Delayed External Cephalic Version in the EECV2 Trial. J Obstet Gynaecol Can. 2016 Mar;38(3):235-245. — http://www.ncbi.nlm.nih.gov/pubmed/27106193